CLINICAL TRIAL: NCT05057715
Title: Phase 1 Trial of Human Chimeric Antigen Receptor Modified T Cells (huCART-meso) Administered in Combination With VCN-01 in Patients With Pancreatic and Serous Epithelial Ovarian Cancer
Brief Title: huCART-meso + VCN-01 in Pancreatic and Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Theriva Biologics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC# 03821, IND #27590
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer; Serous Ovarian Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): Single dose of 3.3x10(12) vp of VCN-01 on Day 0, followed by a single dose of 5x10(7) of huCART-meso cells on Day 14.
  Interventions: Biological: VCN-01; Biological: huCART-meso Cells
- Cohort 2 (Active Comparator): Single dose of 1x10(13) vp of VCN-01 on Day 0, followed by a single dose of 5x10(7) of huCART-meso cells on Day 14.
  Interventions: Biological: VCN-01; Biological: huCART-meso Cells
- Cohort -1 (Active Comparator): In the event that 2 DLTs occur in Cohort 1, then enrollment in Cohort 1 will be stopped and Cohort -1 will be opened for evaluation. Enrolled subjects will receive a single dose of huCART-meso cells on Day 0 followed by a single dose of 3.3x10(12) vp of VCN-01 on Day 14.
  Interventions: Biological: VCN-01; Biological: huCART-meso Cells

INTERVENTIONS:
Biological: VCN-01 — Intravenous administration of VCN-01
Biological: huCART-meso Cells — Intravenous administration of huCART-meso cells

SUMMARY:
This is a Phase I study evaluating the safety and feasibility of lentiviral transduced huCART-meso cells when given in combination with VCN-01 in a 3+3 dose (de)escalation design.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety and feasibility of lentiviral transduced huCART-meso cells when given in combination with VCN-01 in a 3+3 dose (de)escalation design as follows:

* Cohort 1 (N = 3-6): will receive VCN-01 as a single IV infusion of 3.3x1012 vp on Day 0, followed by a single dose of 5x107 huCART-meso cells on Day 14 via IV infusion. This cohort will be evaluated as follows:

  * If 1 DLT/3 subjects occurs, Cohort 1 will be expanded to enroll an additional 3 evaluable subjects.
  * If 0 DLT/3 subjects or 1 DLT/6 subjects, the study will advance to Cohort 2.
* Cohort 2 (N = 3-6): will receive VCN-01 as a single IV infusion of 1x1013 vp on Day 0 followed by a single dose of 5x107 cells huCART-meso cells on Day 14 via IV infusion. This cohort will be evaluated as follows:

  * If 0 DLT/3 subjects or 1 DLT/3 subjects occurs, Cohort 2 will be expanded to enroll an additional 3 evaluable subjects. If 0 DLT/6 subjects or 1 DLT/6 subjects occurs, this dose combination will be identified as the recommended phase 2 dose (RP2D).
  * If 2 DLTs occur at any time, enrollment in this Cohort will be stopped. If less than 6 subjects were infused in Cohort 1 prior to Cohort 2 escalation, additional subjects will be enrolled in Cohort 1to reach a minimum of 6 evaluable subjects.

In the event that 2 DLTs occur in Cohort 1, then enrollment in Cohort 1 will be stopped and Cohort -1 will be opened for evaluation. Cohort -1 will evaluate a different sequence of administration for these two investigational products at the same dose level used in Cohort 1.

• Cohort -1 (N = up to 6): will receive a single dose of 5x107 huCART-meso cells via IV infusions on Day 0 followed by VCN-01 as a single infusion of 3.3x1012 vp on Day 10. Up to 6 subjects will be infused in Cohort -1 unless > 1 DLTs are observed at any time.

The Day 0 infusions of the first two subjects in each cohort will be staggered by at least 42 days from the prior subject's 1st infusion (huCART-meso or VCN-01; depending on the cohort assignment), to allow for the assessment of DLTs and a formal decision regarding cohort progression, expansion, or de-escalation. Subsequent subject infusions within that cohort will be staggered by at least 14 days from the preceding subject's second infusion. Formal DLT assessments will be performed by the Clinical PI and Sponsor Medical Director in accordance with the definition provided in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one of the following diagnoses:

   1. Histologically confirmed unresectable or metastatic pancreatic adenocarcinoma; OR
   2. Persistent or recurrent serous epithelial ovarian cancer
2. Progression or intolerance to at least one prior standard of care chemotherapy for advanced stage disease.
3. Subjects must have measurable disease as defined by RECIST 1.1 criteria.
4. Patients ≥ 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate organ and bone marrow function defined as:

   1. Hemoglobin ≥ 9 g/dL
   2. Platelets ≥ 75,000/µl
   3. PT/INR and PTT ≤ 1.5 x ULN
   4. Bilirubin ≤ 2.0 x ULN
   5. Creatinine ≤ 1.5 x ULN
   6. ALT/AST ≤ 5 x ULN (subjects with liver metastases) or ALT/AST ≤ 2.5 x ULN (subjects without liver metastases)
   7. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
   8. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
7. Provides written informed consent.
8. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in the protocol

Exclusion Criteria:

1. Patients with known CNS metastases
2. Active invasive cancer other than the one of the two cancers targeted by this study. Patients with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder and prostate cancer with PSA level < 1.0) are not excluded.
3. Active hepatitis B or hepatitis C infection.
4. Chronic hepatitis C with a FibroScan score equivalent to fibrosis stage 2 (F2) or greater.
5. Patients with known cirrhosis.
6. Patients with ongoing or active infection.
7. Patients with a known history of Li Fraumeni syndrome or retinoblastoma protein pathway germinal deficiency.
8. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10 mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
9. Planned concurrent treatment with systemic high dose corticosteroids. Patients may be on a stable low dose of steroids (≤ 10mg equivalent of prednisone). Use of inhaled steroids is allowable.
10. Patients requiring supplemental oxygen therapy.
11. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
12. Any clinically significant pericardial effusion, Class II-IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 4) or other cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study. This determination will be made by a cardiologist if cardiac issues are suspected.
13. Pregnant or breastfeeding women.
14. Treatment with a PD-1 or PD-L1 inhibitor, including but not limited to nivolumab, pembrolizumab, atezolizumab, and/or durvalumab, within 2 months prior to eligibility confirmation by a physician-investigator.
15. Patients with significant lung disease as follows:

    1. Patients with radiographic evidence of greater than lobar lymphangitic pulmonary involvement, greater than lobar bronchial wall thickening suggestive of peribronchial lymphatic disease extension, and/or evidence of extensive bilateral parenchymal metastatic burden.
    2. Patients with radiographic and/or clinical evidence of active radiation pneumonitis.
    3. Patients with radiographic evidence of underlying interstitial lung disease, including evidence of unresolved drug toxicity from any agent (e.g. chemotherapy, targeted agents, amiodarone, nitrofurantoin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2038-09 (Estimated); Study Completion 2038-09 (Estimated)

PRIMARY OUTCOMES:
Type, frequency, severity, and attribution of AEs/SAEs as assessed by CTCAE v 5.0 | 2 years
Occurrence of dose-limiting toxicities. | 2 years

SECONDARY OUTCOMES:
Proportion of subjects enrolled who receive one or both of the intended study infusions | 2 years
Overall Response Rate (ORR) | 15 years
Best Overall Response (BOR) | 15 years
Duration of Response (DOR) | 15 years
Progression Free Survival (PFS) | 15 years
Overall Survival (OS) | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Janos L. Tanyi, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided